CLINICAL TRIAL: NCT05041569
Title: Description of Lymphatic Damage in Encephalic Venous Thrombosis and Strictures in MRI a Reverse-recovery Sequence: a Pilot Study
Acronym: ALTREVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JSY_2021_12
Record Dates: First submitted 2021-07-15; First posted 2021-09-13 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Description of Local Modifications of Lymph Nodes or Bundles With the FABIR Sequence in MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI sequences — perform additional sequences added by research

SUMMARY:
Inclusion (J0):

* Information
* Verification of inclusion and non-inclusion criteria
* Collection of consent
* MRI examination with injection of contrast product as part of the treatment comprising the sequences:

T1 TFE 1.0 iso 3D FLAIR injected Injected elliptical venous angiography 0.4mm iso or less 3D SWIp multiecho 3D T1 injected FABIR iso without injection (added as part of care in case of suspected ASH or meningitis) FLAIR 1.0 without injection (added as part of care for suspected ASH or meningitis) T2 BFFE XD (added by search) FABIR iso injected (added by research) 3D PD T1 0.55 MSDE iso injected (added by research)

Clinical information (SRM on inclusion, on discharge and at 3 months and recurrence within the year) will be collected from the patient's medical file

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Performing an MRI injected as part of care for one of the following reasons:
* suspicion of pathology likely to be associated with narrowing or obstruction of one or more venous sinuses (cerebral thrombophlebitis, tissue damage with venous extension, idiopathic HIC
* venous narrowing or obstruction proven by one of the above pathologies, requiring as part of routine care an injected MRI (search for impact, monitoring, pre-therapeutic assessment or prognosis)
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Absolute contraindication to MRI
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presenting for imaging as part of their treatment
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Using a new MRI sequence for the detection of lymph nods | 1 DAY
  Inversion recovery pulse sequences in MRI will be used to detect lymph nods.

CONTACTS AND LOCATIONS:
Locations (1):
- Hhopital fondation adolphe de rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No